CLINICAL TRIAL: NCT01974921
Title: Study of Physiopathological Mechanisms and Results of Treatment With Bronchial Thermoplasty in Severe Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIBSP-TER-2013-70
Record Dates: First submitted 2013-10-22; First posted 2013-11-04 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Thermoplasty; Bronchial smooth muscle
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bronchial thermoplasty (Experimental): ALAIR Catheter. Radiofrequency system.
  Interventions: Device: ALAIR Catheter. Radiofrequency system.

INTERVENTIONS:
Device: ALAIR Catheter. Radiofrequency system. — Radiofrequency with Alair Catheter trhough flexible bronchoscopy in three different sessions (right lower lobe, left lower lobe, both upper lobes).

SUMMARY:
The purpose of this study is to evaluate clinical and histological response to bronchial thermoplasty in severe asthma patients.

DETAILED DESCRIPTION:
Bronchial thermoplasty is a new therapeutic tool for severe and uncontrolled asthma patients. Clinical trials have demonstrated clinical benefits regarding quality of life and exacerbations. Animal models suggested the reduction of bronchial smooth muscle as the principal responsible for the clinical benefits observed in asthma patients treated in the clinical trials, although there is little information about its mechanism of action, and limited to a very small number of case reports. Given that the mechanism of action of bronchial thermoplasty is still not well understood, we proposed a biological study in asthma patients treated with bronchial thermoplasty with the purpose to analyze changes in inflammatory markers and histological samples, as well as its correlation with clinical outcomes in real practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years old.
* Severe persistent asthma according to GINA.
* Inhaled corticosteroids and long-acting ß2 agonist (LABA).
* Other medications for asthma, as oral corticosteroids, anti-IgE, theofiline, etc. are also acceptable.
* Asthma Quality of Life Questionnaire (AQLQ) < 7
* Asthma Control Test (ACT) < 19
* ≥ 2 exacerbations in last year

Exclusion Criteria:

* History of cigarette smoking with > 15 pack/years.
* Other respiratory diseases.
* Comorbidity that can justify the symptoms of the patients.
* Life-threating unstable asthma.
* Any contraindication to perform a bronchoscopy (respiratory insufficiency, coagulation abnormalities, allergy to sedative drugs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Bronchial smooth muscle. | Change from baseline in bronchial smooth muscle at 6 months post-treatment..

SECONDARY OUTCOMES:
Questionnaire of Quality of life (AQLQ) | Change from baseline in AQLQ at 6 months post-treatment.
Questionnaire of asthma control (ACT) | Change from baseline in ACT at 6 months post-treatment.
Number of exacerbations | Change from baseline in number of exacerbations at 6 months post-treatment.
Number of hospitalizations | Change from baseline in number of hospitalizations at 6 months post-treatment.
Respiratory function | Change from baseline in respiratory function at 6 months post-treatment.
Radiological findings (thorax HRCT scan) | Change from baseline in radiological findings at 6 months post-treatment.
Inflammatory markers | Change from baseline in biological inflammatory markers at 6 months post-treatment.
  FeNO eNOSE Bronchial biopsies Sputum Serum

CONTACTS AND LOCATIONS:
Overall Officials: Alfons Torrego, M.D., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain